CLINICAL TRIAL: NCT04299555
Title: Assessment of Fears of Patients Standing at the Operating Block
Status: Completed | Type: Observational
Sponsor: Ch Mont de Marsan (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-Ao1820-55
Record Dates: First submitted 2019-11-15; First posted 2020-03-06 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Anxiety and Fear
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The term "outpatient" refers to all the medical, organizational and administrative care that allows the patient to leave the same day the structure where the ambulatory procedure was performed. The usual rule for patients undergoing endoscopic surgery or surgery under general anesthesia is to transport them to the endoscopy or operating room lying on a stretcher, even if they can walk independently.

In recent years, the procedure of bringing the patient standing in the operating room seems to have many advantages. It is readily accepted by patients and may even lessen their anxiety.

Nevertheless, reluctance and fears are sometimes expressed by patients who do not know this new procedure. Our team has introduced this procedure for patients admitted to the ambulatory hospitalization sector and to join the endoscopy sector.

The aim of our work is therefore to objectify the fears expressed by patients who have to go to the endoscopy room before general anesthesia and to evaluate their progress after endoscopy

DETAILED DESCRIPTION:
Nowadays, the procedure of the patient standing in the operating room or in endoscopy has become frequent in the outpatient management of patients. Indeed the advantages are numerous: better fluidity of the patient circuits to the block, reduction of the stress of the operated one etc. Yet some patients might experience fears.

Thus, in order to improve our practice, we want to take into account your experience with this innovative procedure.

To determine patients' fears concerning their endoscopic standing before general anesthesia and to evaluate their evolution after this first experience

After your installation in the preoperative area, we submit a questionnaire that corresponds to the first part of the document and then accompanied by a hospital agent you will walk towards the entrance to the endoscopy room. These questions are about your possible fears and your degree of anxiety.

After an endoscopy under general anesthesia, you will be taken back to your stretcher room where you will complete the second part of the questionnaire which deals with the same topics as the questions asked before the endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* To be adult (18 years minimum)
* Have a good understanding of the French language
* A diagnosis requiring an endoscopic act.
* Being eligible for outpatient care during anesthesia consultation (ASA I-II and ASA III balanced, good preoperative mobility, understanding pre and postoperative instructions, ability to observe treatments, acceptable housing and hygiene conditions , access to a telephone, journey <1h for the first night).
* Have never been brought before to the operating room or standing endoscopy
* collection of the patient's non-opposition.

Exclusion Criteria:

* refused patient
* Patients with reduced mobility preoperatively
* patient under tutorship or curatorship

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: any patient presenting at the block and corresponding to the criteria over a period of 3 months
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-12-29 (Actual); Study Completion 2018-12-29 (Actual)

PRIMARY OUTCOMES:
determine and assess the fears of the patients who have never been transported to the OR by walking and to reassess their fears after their first experience (Before and after anesthesia) | before anesthesia and after anesthesia, an average of 1 day
  determine the fears expressed by patients who have to go to the endoscopy room before general anesthesia and to evaluate their change after endoscopy with a simple numerical rating scale from 0 to 10 for 5 items. This numerical rating scale is completed by patient at two timepoint: before and after anesthesia. Value 0 corresponding to any fear to value 10 corresponding to maximal fear.

SECONDARY OUTCOMES:
determine the factors associated to these fears (Before and after anesthesia) | before anesthesia and after anesthesia, an average of 1 day
  determine the factors associated to these fears of the patients who have to go to the endoscopy room before general anesthesia and to evaluate their change after endoscopy with a simple numerical rating scale from 0 to 10. This numerical rating scale is completed by patient at two timepoint: before and after anesthesia. Value 0 corresponding to any fear to value 10 corresponding to maximal fear.
determine the anxiety (Before and after anesthesia) | before anesthesia and after anesthesia, an average of 1 day
  evaluate their change of anxiety item before and after endoscopy with a simple numerical rating scale from 0 to 10. This numerical rating scale is completed by patient at two timepoint: before and after anesthesia. Value 0 corresponding to any anxiety to value 10 corresponding to very strong anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Karam SAMII, MD, Principal Investigator — CH de Mont de Marsan
Locations (1):
- centre hospitalier Dax, Dax, France